CLINICAL TRIAL: NCT04692831
Title: Imaging of HER2-expressing Cancer With Site-Specifically Labeled 89Zr-ss-Pertuzumab
Brief Title: Testing a New Imaging Agent to Identify Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-275
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HER-2 Positive Malignant Carcinoma of Breast; HER-2 Protein Overexpression; HER2-positive Metastatic Breast Cancer
Keywords: HER-2 Positive Malignant Carcinoma of Breast; HER-2 Protein Overexpression; HER2-positive Metastatic Breast Cancer; 3+ HER2 IHC; 2+ HER2 IHC; 20-275; Memorial Sloan Kettering Cancer Center; HER2-positive primary malignancy; Zr-ss-Pertuzumab

STUDY DESIGN:
Intervention Model Description: This protocol will perform a first-in-human imaging trial of 89Zr-ss-pertuzumab.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HER2-positive malignancy (Experimental): Participants will have a diagnosis of HER2-positive malignancy
  Interventions: Combination Product: 89Zr-ss-pertuzumab PET/CT
- HER2-low malignancy (Experimental): Participants will have a diagnosis of HER2-low malignancy
  Interventions: Combination Product: 89Zr-ss-pertuzumab PET/CT

INTERVENTIONS:
Combination Product: 89Zr-ss-pertuzumab PET/CT — Patients will receive 89Zr-ss-pertuzumab. 89Zr-ss-pertuzumab PET/CT images will be reconstructed using iterative reconstruction and displayed in multiplanar reconstruction. In the event that 89Zr-ss-pertuzumab is unavailable, randomly labelled 89Zr-pertuzumab PET will be allowed to make HER2 PET imaging available for our patients. Once 89Zr-ss-pertuzumab is available, then patients will be imaged with 89Zr-ss-pertuzumab and randomly labelled 89Zr-pertuzumab will no longer be used.

SUMMARY:
The purpose of this study is to see whether 89Zr-ss-pertuzumab is safe in people with HER2+ cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven HER2-positive or HER2-low primary malignancy or metastatic disease

Note: HER2 positivity is defined according to American Society of Clinical Oncology guidelines or ERBB2 amplification on next generation sequencing Note: HER2-low is defined as low HER2 expression, with immunohistochemistry (IHC) 1+ or IHC 2+ and in situ hybridization [ISH]-negative, including FISH.

* Biopsy proven primary malignancy or metastatic disease
* At least one malignant lesion on CT, MR, or FDG PET/CT within 60 days of protocol enrollment
* Age 18 years or greater
* ECOG performance of 0-2

Exclusion Criteria:

* Creatinine > 2 times normal limit (obtained with 8 weeks of enrollment)
* AST/ALT > 2 times normal limit (obtained with 8 weeks of enrollment)
* Life expectancy < 3 months
* Pregnancy or lactation
* Patients who cannot undergo PET/CT due to weight limits (over 450 pounds)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate clinical safety of 89Zr-ss-pertuzumab | Up to 20 months
  CTCAE Version 5 will be utilized for toxicity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Somali Gavane, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - PATTY AND GEORGE HOAG CANCER CENTER (Data or Specimen Analysis Only), Newport Beach, California
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Yeh R, O'Donoghue JA, Jayaprakasam VS, Mauguen A, Min R, Park S, Brockway JP, Bromberg JF, Zhi WI, Robson ME, Sanford R, Modi S, Agnew BJ, Lyashchenko SK, Lewis JS, Ulaner GA, Zeglis BM. First-in-Human Evaluation of Site-Specifically Labeled 89Zr-Pertuzumab in Patients with HER2-Positive Breast Cancer. J Nucl Med. 2024 Mar 1;65(3):386-393. doi: 10.2967/jnumed.123.266392. PMID 38272704
- [Derived] Zeglis BM, Lewis JS. Click Here for Better Chemistry. N Engl J Med. 2022 Dec 15;387(24):2291-2293. doi: 10.1056/NEJMcibr2213596. Epub 2022 Nov 30. No abstract available. PMID 36449446
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04692831/ICF_000.pdf